CLINICAL TRIAL: NCT04880083
Title: Feeding Tolerance and Gut Maturation of Infants Consuming a Formula Rich in Glycoprotein: A Single-arm, Open-label, Prospective Interventional Study Including a Breastfed Reference Group
Brief Title: Feeding Tolerance and Gut Maturation of Infants Consuming a Formula Rich in Glycoprotein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Medrio, Inc (Unknown); SAS Institute (Industry); Veeva Systems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20.15.INF
Record Dates: First submitted 2021-01-11; First posted 2021-05-10 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Digestion; Gut Microbiota
Keywords: gut tolerance; gut microbiota; gut immunity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formula-Fed (FF) Group (Experimental): Subjects will be fed commercial bovine milk-based, whey-predominant, α-lactalbumin-enriched term formula with high sn-2 palmitate fat blend, supplemented with oligofructose for 6 weeks.
  Interventions: Dietary Supplement: Commercially Available Starter Infant Formula
- Breast-Fed (BF) Group (No Intervention): Subjects will continue exclusive/ predominant breastfeeding for 6 weeks. Breastmilk may be consumed directly from the breast or breast milk may be expressed and fed through infant feeding bottle.

INTERVENTIONS:
Dietary Supplement: Commercially Available Starter Infant Formula — Study formula is provided in powder form and will be administered orally, ad libitum, via an infant feeding bottle and the volume of formula offered to the infant will be guided by the recommended feeding table for the age group or by physician recommendation. The amount consumed by the infant will vary by each infant's weight and appetite.
  Arms: Formula-Fed (FF) Group

SUMMARY:
This is a non-randomized, single-arm, open-label, prospective interventional study using a commercially available starter infant formula in healthy term formula-fed infants with a parallel group of healthy term breast-fed infants as reference group. Approximately 120 male and female infants (60 per group) who are 3-28 days old and are exclusively or predominately formula-feeding or breastfeeding will be enrolled.

DETAILED DESCRIPTION:
Breastmilk contains an abundance of structurally diverse compounds having important physiologic roles. These include glycoproteins which are biologically active and involved in infant gut, immune and brain development (Jiang and Lönnerdal 2016).

The overall purpose of this study is to study the effectiveness of a term infant formula rich in glycoprotein (formula-fed group) on gastrointestinal tolerance, and gastrointestinal health in healthy term infants compared to a breast-fed reference group. We hypothesize that there will be comparable gastrointestinal tolerance in formula-fed and breast-fed and that fecal bifidobacteria changes in early infancy in the formula-fed group are similar to that of breast-fed infants.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of personally signed and dated informed consent document indicating that the infant's parent(s)/ legally accepted representatives LAR have been informed of all pertinent aspects of the study.
2. Infants whose parent(s)/LAR have reached the legal age of majority in the countries where the study is conducted.
3. Infants whose parent(s)/LAR are willing and able to comply with scheduled visits, and the requirements of the study protocol.
4. Infants whose parent(s)/LAR can be contacted directly by telephone throughout the study.
5. Infants whose parent(s)/LAR have a working freezer.
6. Infants must meet all the following inclusion criteria to be eligible for enrolment into the study:

   * Healthy term infant (37-42 weeks of gestation).
   * At enrolment visit, post-natal age 3-28 days (date of birth = day 0)
   * Birth weight ≥ 2500g and ≤ 4500g.
   * Formula-fed infants only: Infants must predominantly consume and tolerate a standard cow's milk infant formula prior to enrolment and their parent(s)/LAR must have independently elected, before enrolment, not to exclusively breastfeed. Predominantly formula feeding means that the infant's predominant source of nourishment has been formula. Specifically, infants are fed with formula for at least 75% of total milk feeds per day.
   * Breastfed infants only: Infants must have been predominantly breastfed since birth, and their parent(s)/LAR must have made the decision to continue predominant breastfeeding for the duration of the study. Predominant breastfeeding allows infants to be mix fed with breastmilk and other milks. It means that the infant's predominant source of nourishment has been breastmilk. Specifically, infants are fed with breast milk for at least 75% of total milk feeds per day.

Exclusion Criteria:

1. Infants with conditions requiring infant feedings other than those specified in the protocol.
2. Infants receiving complementary foods or liquids defined as 4 or more teaspoons per day or approximately 20 g per day of complementary foods or liquids at or prior to enrollment.
3. Infants who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   * Evidence of major congenital malformations (e.g., cleft palate, extremity malformation).
   * Documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis).
   * Previous or ongoing severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigator, would make the infant inappropriate for entry into the study.
4. Infants who are presently receiving or have received prior to enrollment probiotic supplements or any of the following: medication(s) or supplement(s) which are known or suspected to affect the following: fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes); stool characteristics and microbiota (e.g., oral and systemic antibiotics, glycerin suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose); growth (e.g. insulin or growth hormone); gastric acid secretion.
5. Currently participating or having participated in another clinical trial since birth.
6. Subjects or subjects' parent(s) or legal representative who are not willing and not able to comply with scheduled visits and the requirements of the study protocol.

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Overall gastrointestinal (GI) tolerance | Day 39-45
  Compare the overall gastrointestinal (GI) tolerance between the formula-fed and the breast-fed infants from enrolment to 6 weeks of intervention.
  Assessed through the IGSQ-13 (Infant Gastrointestinal Symptoms Questionnaire). The IGSQ-13, consisting of 13 questions, is a retrospective, standardized, validated, questionnaire of GI symptoms and related behaviors that the infant experienced over the past week from a parent's perspective. Overall GI tolerance is assessed from the IGSQ index score, computed from the 13 questions. Possible scores range from 13 - 65, with lower scores representing lower overall GI burden.

SECONDARY OUTCOMES:
Change in Bifidobacteria abundance | Day 1, Day 36-44
  Change in Bifidobacteria abundance from baseline to be measured in the stool samples collected.
Fecal microbiota | Day 1, Day 36-44
  Overall fecal microbiota composition and diversity and community type. Diversity will include relative abundance of beneficial and pathogenic bacteria species (such as beneficial bifidobacteria diversity). To be measured in stool samples collected.
Fecal metabolism | Day 1, Day 36-44
  To be measured in stool samples collected. The metabolic profile consist of pH and organic acids (such as but not restricted to acetate, lactate, butyrate, and propionate), analyzed using HPLC.
GI immunity assessed from fecal markers | Day 1, Day 36-44
  To be measured in stool samples collected. Fecal markers include fecal secretory IgA measured by ELISA. Cytokine profile (such as, but not restricted to: IL-1ra, IL1-alpha, IL-1beta, IL-6, IFN-gamma, and TNF-alpha) measured by multiplex assays. OPV-specific IgA measured by ELISA.
GI maturation assessed from fecal markers | Day 1, Day 36-44
  To be measured in stool samples collected. Includes fecal markers of GI health and maturation assessed by ELISA, such as but not restricted to α-1-antitrypsin and lipocalin.
Stool characteristics: Stool frequency | Day 0, Day 36-44
  Stool frequency using the 1-day and 3-day Stooling and Milk Intake Diary.
Stool characteristics: Difficulty in passing stool | Day 0, Day 36-44
  Difficulty in passing stool using the 1-day and 3-day Stooling and Milk Intake Diary.
Stool characteristics: Stool consistency | Day 0, Day 36-44
  Stool consistency using a 5-point scale in the 1-day and 3-day Stooling and Milk Intake Diary.
GI-related behaviors: Stooling | Day 0, Day 39-45
  Baby bowel movements using the individual IGSQ (Infant Gastrointestinal Symptoms Questionnaire) questions.
GI-related behaviors: Incidence of spitting-up | Day 0, Day 39-45
  Incidence of spitting-up using the individual IGSQ (Infant Gastrointestinal Symptoms Questionnaire) questions.
GI-related behaviors: Crying time | Day 0, Day 39-45
  Baby crying time using the individual IGSQ (Infant Gastrointestinal Symptoms Questionnaire) questions.
GI-related behaviors: Fussiness | Day 0, Day 39-45
  Baby fussiness using the individual IGSQ (Infant Gastrointestinal Symptoms Questionnaire) questions.
GI-related behaviors: Incidence of flatulence | Day 0, Day 39-45
  Flatulence using the individual IGSQ (Infant Gastrointestinal Symptoms Questionnaire) questions.
Milk intake (Breast-Fed infants) | Day 0, Day 36-44
  Total number of feedings using the 1-day and 3-day Stooling and Milk Intake Diary.
Milk intake (Formula-Fed infants) | Day 0, Day 36-44
  Total number of feedings and total quantity of milk consumed for every formula-feeding using the 1-day and 3-day Stooling and Milk Intake Diary.
Infant quality of life | Day 0, Day 39-45
  Assessed from the Infant Quality of Life Questionnaire (IQI). The IQI is a short, age-appropriate, and relevant tool that assesses 8 health-related domains in infants up to 1 year. The domains are sleeping, feeding, breathing, stooling, mood, skin, interaction and other health problems.
Growth: Weight of the infant | Day 0, Day 39-45
  Weight in grams and corresponding weight-for-age Z-score according to the WHO growth standards.
Growth: Length of the infant | Day 0, Day 39-45
  Length in centimeters and corresponding length-for-age Z-score according to the WHO growth standards.
Growth: Weight-for-length of the infant | Day 0, Day 39-45
  Corresponding weight-for-length Z-score according to the WHO growth standards.
Growth: Head circumference of the infant | Day 0, Day 39-45
  Head circumference in centimeters and corresponding head-circumference-for-age Z-score according to the WHO growth standards.
Growth: Body mass index (BMI) of the infant | Day 0, Day 39-45
  Weight and height will be combined to report the BMI (kg/m2) and corresponding BMI-for-age Z-score according to the WHO growth standards.
Safety assessment: Infant illness | Day 0 through 14 days after Day 39-45
  As part of the standard adverse events (AEs) reporting for safety assessment.
Safety assessment: Infection outcomes | Day 0 through 14 days after Day 39-45
  As part of the standard adverse events (AEs) reporting for safety assessment.
Safety assessment: Medication use | Day 0 through 14 days after Day 39-45
  As part of the standard adverse events (AEs) reporting for safety assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Principal Investigator — Shanghai Institute for Pediatric Research at Xinhua Hospital, Shanghai Jiao Tong University
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, China